CLINICAL TRIAL: NCT00393913
Title: Relating Sleep Disordered Breathing to Daytime Function
Brief Title: Evaluating the Relationship Between Sleep-Disordered Breathing and Daytime Alertness
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1357; R01HL081310-01A1 (NIH)
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea; Sleep-Disordered Breathing; Snoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Snoring | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Continuous Positive Airway Pressure (CPAP): Participants will use a CPAP machine if they are found to have sleep apnea.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Positive airway pressure delivered via a nasal mask titrated to a therapeutic level to eliminate all sleep disordered breathing to be used every night for 4-6 weeks.

SUMMARY:
Obstructive sleep apnea (OSA) is a serious sleep disorder in which a person repeatedly stops breathing, or experiences shallow breathing for short periods of time during sleep. Daytime sleepiness is a common symptom of OSA and may affect an individual's level of alertness throughout the day. The primary purpose of this study is to evaluate the relationship between the severity of sleep-disordered breathing and levels of daytime alertness at baseline (untreated state) in a group of subjects with and without sleep apnea. In addition the change in daytime sleepiness in subjects with sleep apnea being treated with a continuous positive airway pressure (CPAP) machine, a common treatment for OSA will also be assessed.

DETAILED DESCRIPTION:
Individuals with OSA can experience up to 300 sleep disruptions each night, which may result in excessive daytime sleepiness (EDS), one of the most common symptoms of OSA. EDS can have serious consequences, including motor vehicle accidents, poor school performance, and work-related accidents and performance issues. The most common treatment for OSA is CPAP therapy. This involves wearing a mask over the nose while sleeping; air then flows through the mask into the nose to maintain a level of pressure that keeps the breathing passages open. CPAP therapy typically results in fewer sleep and breathing disruptions during the night, which may increase an individual's alertness levels during the day. The purpose of this study is to evaluate the relationship between severity of sleep-disordered breathing and daytime alertness levels in adults with and withoutout symptoms of OSA.

This study will involve three to five study visits over a 2- to 3-month period. During the first 3 days, participants will record their sleep habits in a diary and will wear a device that measures breathing, oxygen levels, and sleep position. All participants will then take part in a 1-night inpatient stay at the sleep center lab during which brain, eye, muscle, heart, and breathing activity will be monitored. Participants with a confirmed diagnosis of OSA will stay at the sleep lab one additional night for observation while using a CPAP machine. The following day, tests to measure alertness, ease of falling asleep, and sleepiness levels will be administered. Participants will then use the CPAP machine at home for 4-6 weeks; each machine will be set at an appropriate level for the participant, and will record breathing patterns and pressure. Participants will receive weekly phone calls for monitoring purposes. At the end of Week 4, participants will return to the sleep lab for one additional night of CPAP monitoring, followed by alertness and sleep testing. Those with severe OSA will use the CPAP machine at a newly adjusted level for 5 additional days and return for repeat testing. All participants who have been compliant with CPAP will return to the lab for overnight sleep testing without the CPAP machine and for alertness testing.

ELIGIBILITY:
Inclusion Criteria:

* Experiences symptoms of OSA, including snoring and sleepiness
* Stable medical history with no change in medications that could affect sleepiness

Exclusion Criteria:

* Suspected diagnosis of a sleep disorder other than OSA (i.e., periodic leg movements, narcolepsy, insomnia, central sleep apnea, sleep hypoventilation syndrome)
* Medically unstable health conditions (e.g., heart attack, congestive heart failure)
* Use of psychotropic medications that cause sedation in the 3 months prior to study entry
* Recent or confirmed history of recreational drug use or alcohol abuse
* Pregnant
* Inability to communicate verbally, write, or read
* Visual, hearing, or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects coming to the NYU sleep center with complaints of sleep disordered breathing and normal controls.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2006-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indu Ayappa, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Sleep Disorders Center, New York, New York, United States

REFERENCES:
- [Result] Somiah M, Taxin Z, Keating J, Mooney AM, Norman RG, Rapoport DM, Ayappa I. Sleep quality, short-term and long-term CPAP adherence. J Clin Sleep Med. 2012 Oct 15;8(5):489-500. doi: 10.5664/jcsm.2138. PMID 23066359
- [Result] Young LR, Taxin ZH, Norman RG, Walsleben JA, Rapoport DM, Ayappa I. Response to CPAP withdrawal in patients with mild versus severe obstructive sleep apnea/hypopnea syndrome. Sleep. 2013 Mar 1;36(3):405-12. doi: 10.5665/sleep.2460. PMID 23449493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Normal volunteers and patients with symptoms of sleep apnea evaluated at the NYU sleep disorders center.
Pre-assignment Details: Subjects with sleep disorders other than sleep apnea were not included for initial assessment of the effect of sleep apnea severity to daytime function.
Groups:
- CPAP: All participants with sleep apnea will use a CPAP machine for treatment of sleep apnea.
Period: Initial Assessment
Arm/Group | CPAP
Started | 144
Completed | 107
Not Completed | 37
Not completed — diagnosed with other sleep disorder | 21
Not completed — Withdrawal by Subject | 16
Period: CPAP
Arm/Group | CPAP
Started | 100 (Excludes normal volunteers without OSA)
Completed | 93
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — TEchnical problem with CPAP | 3
Period: CPAP Withdrawal
Arm/Group | CPAP
Started | 42 (Includes only subjects with good CPAP adherence)
CPAP Compliance | 42 (Only subjects with sufficient CPAP complaince (>4 hrs/night) were included.)
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 107 total, with 87 subjects with sleep apnea and 20 without sleep apnea.
Groups:
- Sleep Apnea Assessment: All participants were assigned to a single Arm (and received the intervention based on whether they had sleep apnea). Participants with sleep apnea used the CPAP machine for 4 to 6 weeks every night and then returned to the sleep laboratory for assessment of daytime function. Those without sleep apnea will have the initial assessment but then will not receive the intervention.
Arm/Group | Sleep Apnea Assessment
Number analyzed (Participants) | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 69
Region of Enrollment [Number; unit: participants]
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Subjective Sleepiness
Description: Measured using the Epworth sleepiness scale (ESS). The Epworth sleepiness scale is used in the assessment of daytime sleepiness and measures the general level of sleepiness.The ESS presents the subject with eight situations and asks how likely they are to fall asleep (0= never, 1 =slight chance of dozing, 2= moderate chance of dozing and 3 =high chance of dozing) in these situations. The sum of the 8 answers is used as the score and ranges from 0 (not sleepy) to 24 (extremely sleepy), and a score of greater than 10 is an indication that a person may be excessively sleepy.
Time Frame: Baseline, CPAP( 4 -6 weeks), Off CPAP ( 2 nights)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sleep Apnea: All participants with obstructive sleep apnea (and no other sleep disorder) and subjects without sleep apnea.
Arm/Group | Sleep Apnea
Number analyzed (Participants) | 107
units on a scale
  Baseline ESS | 11.8 (5.6)
  CPAP ESS | 10.2 (5.0)
  CPAP withdrawal ESS | 9.9 (4.6)

2. Primary Outcome: Objective Sleepiness
Description: Multiple Sleep Latency Test (MSLT) measures the latency to sleep onset in minutes. The shorter the latency to sleep the more sleepy the subject.
Time Frame: Measured at baseline, on CPAP (4-6 weeks), CPAP withdrawal (2 nights)
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Continuous Positive Pressure Treatment: All participants with sleep apnea will use a CPAP machine for treatment of sleep apnea.
Arm/Group | Continuous Positive Pressure Treatment
Number analyzed (Participants) | 107
minutes
  Sleep Latency-Baseline | 6.4 (3.7)
  Sleep Latency-CPAP | 5.9 (3.1)
  Sleep Latency-CPAP withdrawal | 7.8 (4.1)

3. Primary Outcome: Vigilance
Description: Vigilance is measured using the psychomotor vigilance task which is a portable reaction time test that is contained in a small, programmable, portable electronic box that requires only a single switch to start. The task consists of responding to a small bright red light stimulus by pressing a response button as soon as the stimulus appears. This stops the stimulus counter and displays the reaction time (RT) in milliseconds for a 2-second period and the task duration is 20 minutes. The subject is instructed to press the button as soon as each stimulus appears in order to keep the reaction time as low as possible. The PVT yields highly informative metrics on the capacity for sustained attention including the frequency of lapses (reaction time > 500 milliseconds). The higher the number of lapses the greater the impairment. Well rested (non-sleepy) subjects have almost no lapses(<2) during the 20min test.
Time Frame: Baseline, CPAP (4-6 weeks), CPAP withdrawal (2 nights)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Lapses
Arm/Group | Continuous Positive Pressure Treatment
Number analyzed (Participants) | 107
Lapses
  Baseline | 5.9 (4.1)
  CPAP | 4.1 (2.6)
  CPAP withdrawal | 6.5 (4.5)

ADVERSE EVENTS:
Arm/Group | Continuous Positive Pressure Treatment
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No